CLINICAL TRIAL: NCT03873987
Title: A Randomized, Open-label, PK and Safety Study to Evaluate the Relative Exposure and Safety of a New Formulation vs the Approved Formulation of a Single 1200 mg IV Dose of ORBACTIV® (Oritavancin) in Subjects Being Treated for ABSSSI
Brief Title: Relative Exposure and Safety Study of Kimyrsa in ABSSSI Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ML-ORI-102
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Acute Bacterial Skin and Skin Structure Infection
MeSH Terms: interventions — oritavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Current Formulation of Oritavancin (Active Comparator): Three single-use vials, each containing 400 mg (1200 mg total) of oritavancin diphosphate (as the free base) and the inactive component mannitol. Oritavancin vials will be reconstituted with SWFI and further diluted in D5W for a total volume of 1000 mL and infused intravenously over 3 hours.
  Interventions: Drug: Current Formulation of Oritavancin
- Kimyrsa (Experimental): A single vial containing 1200 mg of oritavancin, HPβCD, and mannitol. Kimyrsa vials will be reconstituted with SWFI and further diluted with 0.9% sodium chloride for a total volume of 250 mL and infused intravenously over 1 hour.
  Interventions: Drug: Kimyrsa

INTERVENTIONS:
Drug: Current Formulation of Oritavancin — Current formulation of oritavancin (3 hour infusion of 1200 mg in 1000 ml of D5W)
  Other Names: Orbactiv
  Arms: Current Formulation of Oritavancin
Drug: Kimyrsa — New formulation of oritavancin (1 hour infusion of 1200 mg in 250 ml of saline)
  Arms: Kimyrsa

SUMMARY:
This study is being conducted to evaluate the pharmacokinetic (PK) and safety of Kimyrsa versus the approved oritavancin formulation in subjects with acute bacterial skin and skin structure infection (ABSSSI). Kimyrsa adjusts the infusion time, concentration and reconstitution/administration solutions of a single 1200 mg intravenous (IV) infusion of oritavancin

DETAILED DESCRIPTION:
Single IV dose oritavancin (1200 mg) has been approved in the U.S. for the treatment of adult patients with ABSSSI caused or suspected to be caused by Gram-positive microorganisms. The current study is being conducted to evaluate the relative exposure, PK and safety of a new formulation of oritavancin, Kimyrsa, by adjusting infusion time, concentration and reconstitution/administration solutions of a single 1200 mg IV infusion of oritavancin in adult subjects with ABSSSI.

Fifty (50) subjects will be administered the currently approved formulation of oritavancin, using the approved dosing regimen in which Sterile Water for Injection (SWFI) is the reconstituting agent and Dextrose 5% in Water (D5W) is used for further dilution to a total volume of 1000 mL. This formulation will be infused per the approved label over 3 hours. An additional 50 subjects will be administered Kimyrsa which contains hydroxypropyl-β-cyclodextrin (HPβCD). This formulation will be reconstituted with SWFI and further diluted in 0.9% sodium chloride (saline) to a total volume of 250 mL. This formulation will be infused over 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study if they meet all of the following criteria:

1. Subject must be 18 years of age or older, male or female, and of any race.
2. Subject must give written informed consent before initiation of any study-related procedures.
3. Diagnosis of ABSSSI (wound infections, cellulitis/erysipelas, or cutaneous abscess) suspected or confirmed to be caused by a Gram-positive pathogen requiring IV therapy.
4. If female, the subject is surgically sterile, postmenopausal, or, if of childbearing potential, agrees to use at least 2 highly effective methods of birth control (e.g. prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods, abstinence) for the duration of the study until 60 days after study drug administration, or male partner sterilization alone.
5. Subject must express a commitment to comply with all study visits, procedures and requirements for the duration of the study.

Exclusion Criteria

Subjects will be excluded from the study if any of the following exclusion criteria apply prior to randomization:

1. Infections associated with, or in close proximity to, a prosthetic device.
2. Severe sepsis or refractory shock.
3. Known or suspected bacteremia at time of screening.
4. ABSSSI due to or associated with any of the following:

   1. Infections suspected or documented to be caused by only Gram-negative pathogens (i.e., infections acquired during prolonged admission in hospital or long-term care facilities).
   2. Diabetic foot infections (infection extending distal to the malleoli in a subject with diabetes mellitus and peripheral neuropathy and/or vascular insufficiency or any ulceration of their foot).
   3. Concomitant infection at another site not including a secondary ABSSSI lesion (e.g., septic arthritis, endocarditis, osteomyelitis).
   4. Infected burns.
   5. A primary infection secondary to a pre-existing skin disease with associated inflammatory changes such as atopic dermatitis, eczema, or hidradenitis suppurativa.
   6. Decubitus or chronic skin ulcer, or ischemic ulcer due to peripheral vascular disease (arterial or venous).
   7. Any evolving necrotizing process (i.e., necrotizing fasciitis), gangrene or infection suspected or proven to be caused by Clostridium species (e.g., crepitance on examination of the ABSSSI site and/or surrounding tissue(s) or radiographic evidence of subcutaneous gas in proximity to the infection).
   8. Infections known to be caused by an organism resistant to oritavancin.
   9. Catheter site infections.
5. Treatment with investigational medicinal product within 30 days or 5 half-lives, whichever is longer, before enrollment and for the duration of the study.
6. Subjects currently receiving anticoagulant therapy.
7. Known liver function tests (LFTs) ≥ 3 times the upper limit of normal (ULN) or total bilirubin ≥ 2 times ULN.
8. Any medical condition, which in the judgment of the Investigator, might interfere with the pharmacokinetics, distribution, metabolism, or excretion of the study drug.
9. Any planned, major surgical procedure during the study period (Day 15).
10. Subject is the Investigator or his/her deputy, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
11. Known hypersensitivity to oritavancin, glycopeptides or HPβCD.
12. Female subject who has a positive pregnancy test or is breastfeeding.
13. Previous use of oritavancin or anticipated need to use a long acting glycopeptide during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue K Cammarata, MD, Study Director — Melinta Therapeutics, Inc.
Locations (4):
- United States (4):
  - ML-ORI-102 Study Site, Chula Vista, California
  - ML-ORI-102 Study Site, La Mesa, California
  - ML-ORI-102 Study Site, Burr Ridge, Illinois
  - ML-ORI-102 Study Site, Somers Point, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- New Formulation of Oritavancin: A single vial containing 1200 mg of oritavancin, HPβCD, and mannitol. Oritavancin vials will be reconstituted with SWFI and further diluted with 0.9% sodium chloride for a total volume of 250 mL and infused intravenously over 1 hour.
  New Formulation of Oritavancin: New formulation of oritavancin (1 hour infusion of 1200 mg in 250 ml of saline)
Period: Overall Study
Arm/Group | Current Formulation of Oritavancin | New Formulation of Oritavancin
Started | 52 | 50
Completed | 50 | 49
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — staff was unable to start a new IV line | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Current Formulation of Oritavancin | New Formulation of Oritavancin | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (12.1) | 42.1 (12.7) | 44.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 37 | 30 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 21 | 42
  Not Hispanic or Latino | 31 | 29 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 45 | 46 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 50 | 102
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.3 (6) | 29.7 (8.5) | 28.5 (7.4)
Weight [Mean (Standard Deviation); unit: kg] | 80.8 (19.5) | 88.7 (26.9) | 84.7 (23.7)

OUTCOME MEASURES:

1. Primary Outcome: Relative Exposure of AUC of the New Formulation to the Approved Formulation
Description: Relative exposure of AUC of the new formulation to the approved formulation of oritavancin based on area under the plasma concentration-time curve from time zero to 72 hr (AUC0-72)
Time Frame: 72 hours
Population: PK Population: all subjects who have received the full dose of oritavancin and have any valid samples measured for study drug levels
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Groups:
- Orbactiv: Three single-use vials, each containing 400 mg (1200 mg total) of oritavancin diphosphate (as the free base) and the inactive component mannitol. Orbactiv vials were reconstituted with SWFI and further diluted in D5W for a total volume of 1000 mL and infused intravenously over 3 hours.
- Kimrysa: A single vial containing 1200 mg of oritavancin, HPβCD, and mannitol. Kimrysa vial was reconstituted with SWFI and further diluted with 0.9% sodium chloride for a total volume of 250 mL and infused intravenously over 1 hour.
Arm/Group | Orbactiv | Kimrysa
Number analyzed (Participants) | 50 | 50
h*µg/mL | 1470 (39.7) | 1460 (35.1)

2. Primary Outcome: Relative Exposure of AUC of the New Formulation to the Approved Formulation
Description: Relative exposure of AUC of the new formulation to the approved formulation of oritavancin based on area under the plasma concentration-time curve from time zero to 168 hr (AUC0-168).
Time Frame: 168 hours (Day 8)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Orbactiv | Kimrysa
Number analyzed (Participants) | 50 | 50
h*µg/mL | 1760 (41.4) | 1750 (35)

3. Secondary Outcome: Number of Subjects With at Least One Treatment Emergent Adverse Event (TEAE)
Description: Number of subjects with at least one treatment emergent adverse event (TEAE)
Time Frame: 336 hours (Day 15)
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Groups:
- Kimyrsa: A single vial containing 1200 mg of oritavancin, HPβCD, and mannitol. Kimrysa vial was reconstituted with SWFI and further diluted with 0.9% sodium chloride for a total volume of 250 mL and infused intravenously over 1 hour.
Arm/Group | Orbactiv | Kimyrsa
Number analyzed (Participants) | 52 | 50
Participants | 31 | 24

ADVERSE EVENTS:
Time Frame: From the time of study drug initiation to Day 15
Description: Adverse events and serious adverse events will be assessed from the time of study drug administration through Day 15 post administration of oritavancin. AEs will be collected at every subject visit.
Arm/Group | Orbactiv | Kimrysa
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/50
Other Adverse Events (participants affected / at risk) | 31/52 | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orbactiv (N=52) | Kimrysa (N=50)
worsening of left leg cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Orbactiv (N=52) | Kimrysa (N=50)
Hypersensitivity (Immune system disorders) | 2 | 1
Abscess (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 3 | 2
Oral candidiasis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
concussion (Injury, poisoning and procedural complications) | 1 | 0
contusion (Injury, poisoning and procedural complications) | 1 | 0
overdose (Injury, poisoning and procedural complications) | 1 | 0
road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
skin laceration (Injury, poisoning and procedural complications) | 1 | 0
upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
alanine aminotransferase increased (Investigations) | 1 | 0
aspartate aminotransferase increased (Investigations) | 1 | 0
heart rate increased (Investigations) | 0 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
headache (Nervous system disorders) | 0 | 2
presyncope (Nervous system disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 1
diarrhoea (Gastrointestinal disorders) | 5 | 3
nausea (Gastrointestinal disorders) | 3 | 1
toothache (Gastrointestinal disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 2 | 0
chills (General disorders) | 1 | 3
drug withdrawal syndrome (General disorders) | 1 | 0
infusion site extravasation (General disorders) | 1 | 1
pyrexia (General disorders) | 1 | 3
infusion site pain (General disorders) | 0 | 1
infusion site swelling (General disorders) | 1 | 0
oedema (General disorders) | 1 | 0
oedema peripheral (General disorders) | 0 | 1
peripheral swelling (General disorders) | 1 | 0
dysuria (Renal and urinary disorders) | 0 | 1
scrotal oedema (Reproductive system and breast disorders) | 0 | 1
pruritus (Skin and subcutaneous tissue disorders) | 7 | 2
pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 3
red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No such presentation or publication will be initiated by PI until earliest to occur of the following (i) 12 months after the conclusion of the study (ii) publication by the Sponsor or the lead investigator or (iii) written approval is obtained by the Sponsor. PI will provide Sponsor with a draft of any proposed presentation or publication for review at least 45 days in advance of the submission, presentation or publication date.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT03873987/SAP_000.pdf
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03873987/Prot_001.pdf